CLINICAL TRIAL: NCT05739123
Title: Relugolix Pregnancy Registry: An Observational Study of the Safety of Relugolix-Containing Therapy Exposure in Pregnant Women and Their Offspring
Status: Recruiting | Type: Observational
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MVT-601A-002
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Pregnancy Complications; Pregnancy, High Risk
Keywords: Relugolix; Uterine Fibroids; Endometriosis; Pregnancy
MeSH Terms: conditions — Pregnancy Complications; Leiomyoma; Endometriosis | interventions — relugolix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Exposed Cohort: Pregnant women who are exposed to relugolix-containing therapy at any time during pregnancy
  Interventions: Drug: Relugolix-Containing Product
- Unexposed Cohort: Pregnant women with conditions for which relugolix-containing therapy may be prescribed for indications that are approved or under phase 3 development and who are not exposed to relugolix-containing therapy at any time during pregnancy

INTERVENTIONS:
Drug: Relugolix-Containing Product — Any relugolix-containing therapy
  Other Names: TAK-385; T-1331285; RVT-601; MVT-601; MVT-601A; MYFEMBREE
  Groups: Exposed Cohort

SUMMARY:
The Relugolix Pregnancy Registry is a prospective, observational cohort study designed to evaluate the association between relugolix-containing therapy exposure during pregnancy and subsequent maternal, fetal, and infant outcomes. Data will be collected from enrolled pregnant women and the healthcare providers (HCPs) involved in their care or the care of their infants, if applicable.

DETAILED DESCRIPTION:
The outcomes of interest include major congenital malformation (MCM; primary outcome), minor congenital malformation, spontaneous abortion (SAB), stillbirth, elective termination, small for gestational age (SGA), preterm birth, postnatal growth deficiency, and infant developmental deficiency.

Pregnancy outcomes will be assessed throughout pregnancy, with data collection occurring at enrollment, the end of the second trimester, and pregnancy outcome. Infant outcomes will be assessed throughout the infant's first year of life, with active data collection by the registry occurring at 4 and 12 months after delivery. Enrolled pregnant women and the healthcare providers (HCPs) involved in their care or the care of their infants, if applicable, will serve as data reporters to the registry.

The registry is strictly observational; the schedule of office visits and all treatment regimens will be determined by HCPs. Only data that are documented in patients' medical records during the course of medical care will be collected. No additional laboratory tests or HCP assessments will be required as part of this registry.

ELIGIBILITY:
Inclusion Criteria:

* Woman of any age
* Currently or recently pregnant
* Consent to participate
* Authorization for her HCP(s) to provide data to the registry

Cohort 1

* Exposure to at least one dose of relugolix-containing therapy at any time during pregnancy

Cohort 2

* Diagnosis of a condition for which relugolix-containing therapy may be prescribed and who are not exposed to relugolix containing therapy at any time during pregnancy

Exclusion Criteria:

The following will be eligible for enrollment, included in supplementary analyses, but excluded from the analysis population:

* Occurrence of pregnancy outcome prior to first contact with the registry coordination center (retrospectively enrolled)
* Exposure to known teratogens and/or investigational medications during pregnancy
* Lost to follow-up

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will include 2 cohorts of pregnant women: one cohort exposed to relugolix-containing therapy and one cohort of women with conditions for which relugolix-containing therapy may be prescribed and who are not exposed to relugolix-containing therapy.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Major Congenital Malformation (MCM) | Up to 10 years
  Comparison of rate of MCM between cohorts

SECONDARY OUTCOMES:
Minor congenital malformations | Up to 10 years
  Comparison of rate of minor congenital malformations between cohorts
Spontaneous abortion (SAB) | Up to 10 years
  Comparison of rate of SABs between cohorts
Stillbirth | Up to 10 years
  Comparison of rate of stillbirths between cohorts
Elective termination | Up to 10 years
  Comparison of rate of elective terminations between cohorts
Preterm birth | Up to 10 years
  Comparison of rate of preterm births between cohorts
Small for gestational age (SGA) | Up to 10 years
  Comparison of rate of SGA between cohorts
Postnatal growth deficiency | Up to 10 years
  Comparison of rate of postnatal growth deficiency between cohorts
Infant developmental deficiency | Up to 10 years
  Comparison of rate of infant developmental deficiency between cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Wilmington, North Carolina, United States